CLINICAL TRIAL: NCT02912806
Title: The Dartmouth GreenCare Program: Implementation of Shared Decision Making and Patient-reported Outcomes in a Standardized Care Path for Knee Replacement
Brief Title: Dartmouth-Hitchcock GreenCare Registry for Total Knee Replacement
Acronym: GreenCare
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CPHS23310
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: Knee Arthroplasty; Total knee replacement; Knee osteoarthritis; Patient-Outcomes Measurement Program; Surgical Registries; Shared Decision Making; Patient Reported Outcomes; Patient Experience; Cohort Studies
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Total Knee Replacement — Primary total knee arthroplasty for knee osteoarthritis

SUMMARY:
Evolving reimbursement policies are driving health systems to improve quality and efficiency. Transitioning to an electronic health record (EHR) provided Dartmouth-Hitchcock Medical Center (DHMC) an opportunity to redesign staff roles and care path for Total Knee Replacement (TKR). The organization implemented a coordinated team-based care delivery model that integrated real-time measurement of: (1) compliance with trusted guidelines, (2) process of Shared Decision-Making (SdM), and (3) use of Patient-Reported Outcomes (PROs). The investigators present the implementation protocol and data.

DETAILED DESCRIPTION:
Patient-reported outcome measures were completed 1 month preceding TKR and also at 1 and 12 months following surgery. The primary outcome was change in physical function from baseline to 1-year following surgery in the Physical Component Summary (PCS) of the Veterans-Rand (VR-12) Survey. Preoperative measures were: (1) general demographics (patient age, sex, height, weight, body mass index (BMI); (2) treatments tried before surgery; (3) health habits (tobacco use, alcohol use); (4) pre-existing medical conditions (Charlson score); (5) physical exam findings (knee range of motion, knee laxity); (7) lab tests (hemoglobin); and (7) radiographic measures (severity of osteoarthritis on standing x-rays). Secondary outcomes included Physical Score (PS) of the Patient Reported Outcome Measurement Information System Global Survey (PROMIS-10), knee function (Knee Osteoarthritis Outcome Score, KOOS), safety (reoperations, readmissions, emergency visits, and infection) and measures of patient experience (Clinician Group and Hospital Consumer Assessment of Healthcare Providers and Systems).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled TKR
* Osteoarthritis of the knee

Exclusion Criteria:

* previous TKR on the affected knee
* diagnosis other than osteoarthritis
* age less than 18 years
* declined consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduling primary TKR for osteoarthritis of the knee at a regional tertiary care hospital
Sampling Method: Non-Probability Sample
Enrollment: 545 (Actual)
Dates: Start 2013-01; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Health Gain as measured by the change in Physical Component Summary (PCS) Score | 1-year following surgery
  Health Gain from baseline to 12 months (from 300 to 400 days following the date) following surgery, as measured by the change in Physical Score based on standardized US adult population benchmarks for the VR12 survey

SECONDARY OUTCOMES:
Health Gain as measured by the change in Global Physical Health (GPH) | 1-year
  Health Gain from baseline to 12 months following surgery, as measured by the change in Physical Score based on standardized US adult population benchmarks for the PRIOMIS10 survey
Health Gain as measured by the change in Percentile Rank, TKR age and gender matched | 1 year
  Health Gain from baseline to 12 months following surgery, as measured by the change in Physical Score Percentile Rank based on age and gender-matched beta distributions for the Dartmouth TKR population, for the PRIOMIS10 or VR12 survey
Emotional Health | 1 year
  Mental Component Summary (MCS) Score change from baseline to 12 months following surgery, as measured by the change in Mental Score based on standardized US adult population benchmarks for the PRIOMIS10 or VR12 survey
Knee Osteoarthritis Outcome Score (KOOS) | 1 year
  Change in KOOS score from baseline to 12 months following surgery
Reoperation | 3 months
  From 0 to 90 days following the date of surgery
Readmission | 3 months
  From 0 to 90 days following the date of surgery
ER visits after surgery | 3 months
  From 0 to 90 days following the date of surgery
Infection | 3 months
  From 0 to 90 days following the date of surgery
Patient Satisfaction with Hospital | 1 month
  HCAHPS survey in 10% random subsample completed between 20 to 40 days following the date of surgery
Patient Satisfaction with Surgeon | 10 months
  Clinician Group CAHPS survey in 10% random subsample completed between 300 to 400 days following the date of surgery
Cost of care | 3 months
  Episode-based costs for 0 to 90 days following the date of surgery, and also per visit outpatient costs
Length of hospital stay | Acute hospitalization
  Number of days between date of admission and date of discharge
Discharge to home | Acute hospitalization
  Disposition at time of discharge from acute hospitalization
Mortality | 1 year
Range of motion | 90 days
  Knee range of motion measured by a clinician between 60 and 120 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sohail K Mirza, MD, MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center

IPD SHARING:
Plan to Share IPD: Yes
The consented data that has been collected will be stripped of all identifiers and kept as a dataset appropriate for sharing with future researchers for secondary analyses. A Project Proposal form and Data Use Agreement will be required.